CLINICAL TRIAL: NCT01575925
Title: A Phase 1 Multi-Center, Open-Label, Dose-Escalation Study to Determine the Pharmacokinetics and Safety of Pomalidomide When Given in Combination With Low Dose Dexamethasone in Subjects With Relapsed or Refractory Multiple Myeloma and Impaired Renal Function
Brief Title: Study of Pomalidomide to Evaluate the Pharmacokinetics and Safety for Patients With Multiple Myeloma and Impaired Renal Function (POM Renal)
Acronym: POM Renal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CC-4047-MM-008
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Multiple Myeloma; Renal Impairment
Keywords: Pomalidomide for multiple myeloma; renal impairment; multiple myeloma patients with renal impairment; Pomalidomide for patients with renal impairment due to multiple myeloma; Pomalidomide; dexamethasone; RRMM; impaired renal function in multiple myeloma; hemodialysis; dialysis; POM; Pomalyst; MM; severe renal impairment; CrCl ≤ 30 mL/min; Creatinine less than 30; clinical trial in subjects with multiple myeloma with renal impairement
MeSH Terms: conditions — Multiple Myeloma; Renal Insufficiency | interventions — pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4 mg Oral POM + 40 mg Oral DEX (Experimental): Oral POM at 4 mg on days 1-21 of a 28-day cycle, Oral DEX at 40 mg/day (≤ 75 years old) or 20 mg/day (> 75 years old) on days 1, 8, 15 and 22 of a 28-day cycle
  Interventions: Drug: 4 mg Oral POM + 40 mg Oral DEX
- 2 mg Oral POM + 40 mg Oral DEX (Experimental): Oral POM at 2 mg on days 1-21 of a 28-day cycle, Oral DEX at 40 mg/day (≤ 75 years old) or 20 mg/day (> 75 years old) on days 1, 8, 15 and 22 of a 28-day cycle
  Interventions: Drug: 2 mg Oral POM + 40 mg Oral DEX

INTERVENTIONS:
Drug: 4 mg Oral POM + 40 mg Oral DEX
  Other Names: Pomalidomide (POM); Dexamethasone
  Arms: 4 mg Oral POM + 40 mg Oral DEX
Drug: 2 mg Oral POM + 40 mg Oral DEX
  Other Names: Pomalidomide (POM); Dexamethasone
  Arms: 2 mg Oral POM + 40 mg Oral DEX

SUMMARY:
The purpose of this study is to determine the pharmacokinetics (PK) and safety for the combination of pomalidomide (POM) + low-dose dexamethasone (LD- DEX) in subjects with relapsed or refractory Multiple Myeloma (RRMM) and impaired renal function.

DETAILED DESCRIPTION:
The primary objective of the study is to determine the PK and safety for the combination of POM + (LD-DEX) in subjects with RRMM and impaired renal function.

The secondary objective of the study is to evaluate the efficacy of POM + (LD_DEX) in subjects with RRMM and impaired renal function.

This is a 3+3 dose escalation design, with one cohort each for patients with severely impaired renal function patients (CrCl < 30 mL/min) requiring and not requiring dialysis respectively. There will also be one control cohort with normal renal function, these patients will receive 4 mg POM. Dosing will be 21 days out of a 28 day cycle.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Must be ≥ 18 years at the time of signing the informed consent form
2. Must understand and voluntarily sign an informed consent document prior to any study-related assessments/procedures
3. Must be able to adhere to the study visit schedule and other protocol requirements
4. Must have documented diagnosis of relapsed or refractory multiple myeloma and have measurable disease (serum M-protein ≥ 0.5 g/dL or urine M-protein ≥ 200 mg/24 hours)
5. Must have had at least 1 prior anti-myeloma regimen
6. Must have documented progression as per the International Myeloma Working Group uniform response criteria (Durie, 2006) during or after the last anti-myeloma regimen
7. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
8. Females of childbearing potential (FCBP) must agree to utilize two reliable forms of contraception simultaneously or practice complete abstinence from heterosexual contact for at least 28 days before starting study drug, while participating in the study (including dose interruptions), and for at least 28 days after study treatment discontinuation, and must agree to regular pregnancy testing during this timeframe
9. Females must agree to abstain from breastfeeding during study participation and for 28 following discontinuation from study treatment
10. Males must agree to use a latex condom during any sexual contact with FCBP while participating in the study and for 28 days following discontinuation from study treatment, even if he has undergone a successful vasectomy
11. Males must also agree to refrain from donating semen or sperm while on pomalidomide and for 28 days after discontinuation from study treatment
12. All subjects must agree to refrain from donating blood while on study drug and for 28 days after discontinuation from study treatment
13. All subjects must agree not to share medication

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Peripheral neuropathy ≥ Grade 2
2. Non-secretory multiple myeloma
3. Any of the following laboratory abnormalities:

   * Absolute neutrophil count (ANC) < 1,000/µL
   * Platelet count < 75,000/µL
   * Corrected serum calcium > 14 mg/dL (> 3.5 mmol/L)
   * Hemoglobin < 8 g/dL (< 4.9 mmol/L; prior RBC transfusion or recombinant human erythropoietin use is permitted)
   * Serum glutamic oxaloacetic transaminase/aspartate aminotransferase (SGOT/AST) or serum glutamic pyruvic transaminase/alanine aminotransferase (SGPT/ALT) > 3.0 x upper limit of normal (ULN)
   * Serum total bilirubin > 2.0 mg/dL
4. Prior history of malignancies, other than the disease being studied, unless the subject has been free of the malignancy for ≥ 5 years from initiating study treatment, with the following exceptions:

   * Basal cell carcinoma of the skin
   * Squamous cell carcinoma of the skin
   * Carcinoma in situ of the cervix
   * Carcinoma in situ of the breast
   * Incidental histologic finding of prostate cancer (T1a or T1b using the TNM [tumor, nodes, metastasis] clinical staging system).
5. Previous therapy with Pomalidomide
6. Hypersensitivity to thalidomide, lenalidomide, or dexamethasone
7. Rash ≥ Grade 3 during prior thalidomide or lenalidomide therapy
8. Incidence of gastrointestinal disease that may significantly alter the absorption of pomalidomide
9. Subjects with any one of the following:

   * Congestive heart failure (New York Heart Association Class III or IV)
   * Myocardial infarction within 12 months prior to starting study treatment
   * Unstable or poorly controlled angina pectoris, including Prinzmetal variant angina pectoris
10. Subjects who received any of the following within the last 14 days of initiation of study treatment:

    * Plasmapheresis
    * Major surgery (kyphoplasty is not considered major surgery)
    * Radiation therapy (with the exception of radiation therapy to a pathological fracture site to enhance bone healing or to treat post-fracture pain that is refractory to narcotic analgesics)
    * Any anti-myeloma drug therapy
11. Use of any investigational agents within 28 days or 5 half-lives (whichever is longer) of initiating study treatment
12. Subjects with conditions requiring chronic steroid or immunosuppressive treatment, such as rheumatoid arthritis, multiple sclerosis, and lupus, which likely need additional steroid or immunosuppressive treatments in addition to the study treatment. Includes subjects receiving corticosteroids (> 10 mg/day of prednisone or equivalent) within 3 weeks prior to initiating study treatment
13. Subjects unable or unwilling to undergo antithrombotic prophylactic treatment will not be eligible to participate in this study
14. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
15. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subjects from signing the informed consent form
16. Pregnant or breastfeeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2018-08-07 (Actual); Study Completion 2018-08-07 (Actual)

PRIMARY OUTCOMES:
PK-Area under the plasma concentration time curve (AUC) | Up to 24 times over 7 months
  PK-Area under the plasma concentration time curve (AUC)
PK-Time to maximum plasma concentration (Cmax) | 24 times over 7 months
  PK-Time to maximum plasma concentration (Cmax)
PK-Apparent total body clearance (CL/F) | 24 times up to 7 months
  PK-Apparent total body clearance (CL/F)
PK-Renal clearance (CLr) | 24 times over 7 months
  PK-Renal clearance (CLr)
PK-Apparent volume of distribution (V/F) | 24 times over 7 months
  PK-Apparent volume of distribution (V/F)
PK-Effective terminal half-life (T1/2) | 24 times over 7 months
  PK-Effective terminal half-life (T1/2)

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 5 years
  Number of participants with adverse events (AEs)
Number of participants alive | Up to 5 years
  Number of participants alive
Time to response | Up to 5 years
  Time to response
Duration of response | Up to 5 years
  Duration of response

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers-Squibb, Study Director — Bristol-Myers Squibb
Locations (9):
- United States (7):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Ingalls Cancer Research Center, Harvey, Illinois
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Weill Cornell Medical College, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas
- Canada (2):
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - L'Hotel Dieu de Quebec, Québec

REFERENCES:
- [Background] Li Y, Wang X, O'Mara E, Dimopoulos MA, Sonneveld P, Weisel KC, Matous J, Siegel DS, Shah JJ, Kueenburg E, Sternas L, Cavanaugh C, Zaki M, Palmisano M, Zhou S. Population pharmacokinetics of pomalidomide in patients with relapsed or refractory multiple myeloma with various degrees of impaired renal function. Clin Pharmacol. 2017 Nov 8;9:133-145. doi: 10.2147/CPAA.S144606. eCollection 2017. PMID 29184451
- [Background] Kavanaugh A, Gladman DD, Edwards CJ, Schett G, Guerette B, Delev N, Teng L, Paris M, Mease PJ. Long-term experience with apremilast in patients with psoriatic arthritis: 5-year results from a PALACE 1-3 pooled analysis. Arthritis Res Ther. 2019 May 10;21(1):118. doi: 10.1186/s13075-019-1901-3. PMID 31077258
- [Background] Matous J, et al. MM-008 trial: Pharmacokinetics (PK) and tolerability of pomalidomide plus low-dose dexamethasone (POM plus LoDEX) in relapsed/refractory multiple myeloma (RRMM) patients with renal impairment (RI). Presented at: American Society of Clinical Oncology ASCO 2013, May 31-June 4, 2013, Chicago, IL. Abstract No. 8585. JClinOncol 2013;31(suppl 15):8585-8585.